CLINICAL TRIAL: NCT02324647
Title: Structured Evaluation of adRENal Tumors Discovered Incidentally - Prospectively Investigating the Testing Yield
Acronym: SERENDIPITY
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other); Maastricht University Medical Center (Other); UMC Utrecht (Other); Erasmus Medical Center (Other); Martini Hospital Groningen (Other); Canisius-Wilhelmina Hospital (Other); Diakonessenhuis, Utrecht (Other); Isala (Other); Haga Hospital (Other); St. Antonius Hospital (Other); Kennemer Gasthuis (Other); Maxima Medical Center (Other); Medical Center Alkmaar (Other); Frisius Medisch Centrum (Other); Meander Medical Center (Other); Medisch Spectrum Twente (Other); Onze Lieve Vrouwe Gasthuis (Other); Rijnstate Hospital (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Tergooi Hospital (Other); Vlietland Ziekenhuis (Other); Treant ziekenhuis (Unknown); Flevoziekenhuis (Other)
Responsible Party: Sponsor
Other Study IDs: UGroningen; 4799 (Registry Identifier: Nederlands Trial Register)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2023-06

CONDITIONS: Adrenal Incidentaloma; Adrenocortical Carcinoma
Keywords: Urinary steroid profiling; Adrenal incidentaloma; Adrenocortical carcinoma; cost-effectiveness
MeSH Terms: conditions — Adrenal incidentaloma; Adrenocortical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Urine samples and serum or plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Standard diagnostic work-up for adrenal incidentalomas (AI) consists of periodical biochemical analysis and CT-scanning in case the initial work-up does not demonstrate the presence of hormonal hypersecretion or adrenocortical carcinoma (ACC), respectively. The overall aim of this study is to improve the cost-effectiveness of the diagnostic strategy for AI. Cost-effectiveness of urine steroid profiling (USP) will be compared to the standard diagnostic strategy of repeated CT-imaging.

DETAILED DESCRIPTION:
Rationale: Standard diagnostic work-up for adrenal incidentalomas (AI) consists of periodical biochemical analysis and CT-scanning in case the initial work-up does not demonstrate the presence of hormonal hypersecretion or adrenocortical carcinoma (ACC),respectively. With respect to the diagnosis of ACC, the health benefits of this strategy are controversial for the following reasons: a. critical appraisal of literature has revealed a much lower ACC frequency of 1.9% than previously presumed; b. CT sensitivity and specificity are suboptimal; c. risk of unnecessary adrenalectomies; d. exposure to ionising radiation; e. risk of CT contrast reactions (nephropathy, allergic reaction); f. health care related and economical costs. The hypothesis to be tested is that incorporation of a single baseline urinary steroid profiling (USP) into the management algorithm of AI is more cost-effective than a strategy solely based on repeat CT-scanning.

Objective: SERENDIPITY aims to improve the cost-effectiveness of the diagnostic strategy for AI by the application of a single baseline USP. In addition, we aim to examine the psychological impact for patients with AI being currently subjected to repeated laboratory tests and CT-scanning during several years.

Study design: This is a prospective observational multicenter study. Study population: Patients are eligible if they meet the following inclusion criteria: adrenal mass > 1 cm in diameter incidentally discovered during CT or MRI-scanning, performed for reasons other than an evaluation for adrenal disease and age 18 years or older. The exclusion criteria are: extra-adrenal malignancy (i.e. active or past medical history of malignancy, except for basal cell carcinoma), radiologic diagnosis of simple cyst or bilateral adrenal masses, allergy to radiocontrast, renal insufficiency (i.e. eGFR < 30 ml/min/1.73m2), pregnancy or inability to understand written Dutch.

ELIGIBILITY:
Inclusion Criteria:

* discrete adrenal mass > 1 cm in diameter incidentally discovered during CT/MRI-scanning, performed for reasons other than an evaluation for adrenal disease
* detection CT/MRI-scan performed ≤ 4 months ago
* age 18 years or older.

Exclusion Criteria:

* extra-adrenal malignancy (i.e. active or past medical history of malignancy, except for basal cell carcinoma)
* radiologic diagnosis of simple cyst or bilateral adrenal masses
* allergy to radiocontrast
* renal insufficiency (i.e. eGFR < 30 ml/min/1.73m2)
* pregnancy
* adrenal incidentaloma visible on previous (i.e. > 4 months ago) CT/MRI-scan
* inability to understand written Dutch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research population consists of adult patients with a recently discovered adrenal incidentaloma who meet the selection criteria of SERENDIPITY. A total number of 1000 patients will be included. These subjects will be recruited from the group of patients in whom CT/MRI-scanning has been performed with visualization of the adrenal glands (i.e. CT/MRI scans of abdomen and/or chest, as the latter often include imaging of the upper abdominal region).
Sampling Method: Probability Sample
Enrollment: 807 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness | 2 years
  difference in cost-effectiveness of the current management strategy based on repeat CT-scanning to detect ACC among patients with an AI compared with a strategy using a single baseline USP

SECONDARY OUTCOMES:
frequency of ACC among patients with AI at baseline or during follow-up | 2 years
determination of the percentage of AI that meets the criteria of a malignant CT- phenotype at baseline or during follow-up | 2 years
distribution of pathologic diagnosis in surgically removed adrenal glands | 2 years
QoL in patients with an AI at baseline and during follow-up | 2 years
frequency distribution between hormonal hypersecreting and non-functional AI | 2 years
conversion rate from non-functioning AI towards a hypersecreting AI during follow-up | 2 years
costs of diagnostic procedures and surgical interventions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michiel N Kerstens, MD, PhD, Study Director — University Medical Center Groningen; E Buitenwerf, MD, Principal Investigator — University Medical Center Groningen; P.H.L.T. Bisschop, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; E.M.W. Eekhoff, MD, PhD, Principal Investigator — Free University UMC Amsterdam; E.P.M. van der Kleij-Corssmit, MD, PhD, Principal Investigator — Leiden University Medical Center; R.A. Feelders, MD, PhD, Principal Investigator — Erasmus Medical Center; B. Havekes, MD, PhD, Principal Investigator — Maastricht University Medical Center; H.J.L.M Timmers, MD, PhD, Principal Investigator — UMC St Radboud Nijmegen; G.D. Valk, MD, PhD, Principal Investigator — UMC Utrecht; P.H.N. Oomen, MD, PhD, Principal Investigator — medical center leeuwarden; K.M. van Tol, MD, PhD, Principal Investigator — Martini Hospital Groningen; R.S.M.E. Wouters, MD, Principal Investigator — Scheper Hospital; A.A.M. Franken, MD, PhD, Principal Investigator — Isala; J.R. Meinardi, MD, PhD, Principal Investigator — Canisius-Wilhelmina Hospital; R. GrooteVeldman, MD, PhD, Principal Investigator — Medisch Spectrum Twente; P.C. Oldenburg-Ligtenberg, MD, PhD, Principal Investigator — Meander Medical Center; A.F. Muller, MD, PhD, Principal Investigator — Diakonessenhuis, Utrecht; M.O. van Aken, MD, PhD, Principal Investigator — Haga Hospital; W. de Ronde, MD, PhD, Principal Investigator — Kennemer Gasthuis; H.R. Haak, MD, PhD, Principal Investigator — Maxima Medical Center; S. Simsek, MD, PhD, Principal Investigator — Medical Center Alkmaar; I.M.M.J. Wakelkamp, MD, PhD, Principal Investigator — St. Antonius Hospital; I.I.L. Berk-Planken, MD, PhD, Principal Investigator — Vlietland Ziekenhuis; P.S. van Dam, MD, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis; H. de Boer, MD, PhD, Principal Investigator — Rijnstate Hospital; J.J.J. de Sonnaville, MD, PhD, Principal Investigator — Tergooi Hospital; E. Donga, MD, Principal Investigator — St.Elisabeth Hospital; N. Smit, MD, Principal Investigator — Flevoland Hospital
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Grumbach MM, Biller BM, Braunstein GD, Campbell KK, Carney JA, Godley PA, Harris EL, Lee JK, Oertel YC, Posner MC, Schlechte JA, Wieand HS. Management of the clinically inapparent adrenal mass ("incidentaloma"). Ann Intern Med. 2003 Mar 4;138(5):424-9. doi: 10.7326/0003-4819-138-5-200303040-00013. PMID 12614096
- [Background] Young WF Jr. Clinical practice. The incidentally discovered adrenal mass. N Engl J Med. 2007 Feb 8;356(6):601-10. doi: 10.1056/NEJMcp065470. No abstract available. PMID 17287480
- [Background] Nawar R, Aron D. Adrenal incidentalomas -- a continuing management dilemma. Endocr Relat Cancer. 2005 Sep;12(3):585-98. doi: 10.1677/erc.1.00951. PMID 16172193
- [Background] Kievit J, Haak HR. Diagnosis and treatment of adrenal incidentaloma. A cost-effectiveness analysis. Endocrinol Metab Clin North Am. 2000 Mar;29(1):69-90, viii-ix. doi: 10.1016/s0889-8529(05)70117-1. PMID 10732265
- [Background] Cawood TJ, Hunt PJ, O'Shea D, Cole D, Soule S. Recommended evaluation of adrenal incidentalomas is costly, has high false-positive rates and confers a risk of fatal cancer that is similar to the risk of the adrenal lesion becoming malignant; time for a rethink? Eur J Endocrinol. 2009 Oct;161(4):513-27. doi: 10.1530/EJE-09-0234. Epub 2009 May 13. PMID 19439510
- [Background] Johnson PT, Horton KM, Fishman EK. Adrenal mass imaging with multidetector CT: pathologic conditions, pearls, and pitfalls. Radiographics. 2009 Sep-Oct;29(5):1333-51. doi: 10.1148/rg.295095027. PMID 19755599
- [Background] Wolthers BG, Kraan GP. Clinical applications of gas chromatography and gas chromatography-mass spectrometry of steroids. J Chromatogr A. 1999 May 28;843(1-2):247-74. doi: 10.1016/s0021-9673(99)00153-3. PMID 10399855
- [Background] Grondal S, Eriksson B, Hagenas L, Werner S, Curstedt T. Steroid profile in urine: a useful tool in the diagnosis and follow up of adrenocortical carcinoma. Acta Endocrinol (Copenh). 1990 May;122(5):656-63. doi: 10.1530/acta.0.1220656. PMID 2141212
- [Background] Khorram-Manesh A, Ahlman H, Jansson S, Wangberg B, Nilsson O, Jakobsson CE, Eliasson B, Lindstedt S, Tisell LE. Adrenocortical carcinoma: surgery and mitotane for treatment and steroid profiles for follow-up. World J Surg. 1998 Jun;22(6):605-11; discussion 611-2. doi: 10.1007/s002689900442. PMID 9597936
- [Background] Kikuchi E, Yanaihara H, Nakashima J, Homma K, Ohigashi T, Asakura H, Tachibana M, Shibata H, Saruta T, Murai M. Urinary steroid profile in adrenocortical tumors. Biomed Pharmacother. 2000 Jun;54 Suppl 1:194s-197s. doi: 10.1016/s0753-3322(00)80043-8. PMID 10915023
- [Background] Minowada S, Kinoshita K, Hara M, Isurugi K, Uchikawa T, Niijima T. Measurement of urinary steroid profile in patients with adrenal tumor as a screening method for carcinoma. Endocrinol Jpn. 1985 Feb;32(1):29-37. doi: 10.1507/endocrj1954.32.29. PMID 4017973
- [Background] Brazier J, Roberts J, Deverill M. The estimation of a preference-based measure of health from the SF-36. J Health Econ. 2002 Mar;21(2):271-92. doi: 10.1016/s0167-6296(01)00130-8. PMID 11939242
- [Background] Arnaldi G, Boscaro M. Adrenal incidentaloma. Best Pract Res Clin Endocrinol Metab. 2012 Aug;26(4):405-19. doi: 10.1016/j.beem.2011.12.006. Epub 2012 May 22. PMID 22863384